CLINICAL TRIAL: NCT01605617
Title: Prospective Randomized Trial of Percutaneous Tibial Nerve Stimulation (PTNS) Versus PTNS and Fesoterodine Fumarate
Brief Title: Trial of Percutaneous Tibial Nerve Stimulation (PTNS) Versus PTNS and Fesoterodine Fumarate
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment rate, and study patients were removed prior to completion
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey L. Cornella, Professor of Obstetrics-Gynecology, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11-004589
Record Dates: First submitted 2012-05-03; First posted 2012-05-25 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2013-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTNS + fesoterodine fumarate first, then PTNS + placebo (Active Comparator): Participants were to be given Percutaneous Tibial Nerve Stimulation (PTNS) + 4mg of fesoterodine fumarate first for 12 weeks, and followed by 4 weeks of washout followed by 12 weeks of PTNS + placebo.
  Interventions: Drug: Fesoterodine fumarate; Drug: Placebo; Procedure: Percutaneous Tibial Nerve Stimulation (PTNS)
- PTNS + placebo first, then PTNS + fesoterodine fumarate (Placebo Comparator): Participants were to be given Percutaneous Tibial Nerve Stimulation (PTNS) + placebo for 12 weeks followed by 4 weeks of washout followed by 12 weeks of PTNS + 4mg of fesoterodine fumarate
  Interventions: Drug: Fesoterodine fumarate; Drug: Placebo; Procedure: Percutaneous Tibial Nerve Stimulation (PTNS)

INTERVENTIONS:
Drug: Fesoterodine fumarate — PTNS + 4mg of fesoterodine fumarate for 12 weeks
  Other Names: Toviaz
Drug: Placebo — PTNS + placebo for 12 weeks
Procedure: Percutaneous Tibial Nerve Stimulation (PTNS) — PTNS is an FDA-approved procedure for the diagnosis of overactive bladder, given on a weekly basis. Participants will be given PTNS + either 4mg of fesoterodine fumarate or placebo for 12 weeks, and followed by 4 weeks of washout followed by 12 weeks of PTNS + the opposite treatment (placebo or fesoterodine fumarate).

SUMMARY:
The investigators are studying two FDA-approved modalities used to treat overactive bladder to determine if they improve overactive bladder with or without urge incontinence when used together rather than separately, percutaneous tibial nerve stimulation (PTNS) versus PTNS and fesoterodine fumarate.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is described as urinary urgency with or without urge incontinence, usually associated with urinary frequency and nocturia. The primary complaint is a strong desire to void without the ability to postpone micturition. Two treatments used in the treatment of OAB are pharmacotherapy and percutaneous tibial nerve stimulation (PTNS).

Pharmacotherapy for OAB is based on medications that block the muscarinic receptors of the detrusor muscle. These particular receptors are not unique to the bladder, however, and patients complain of bothersome side effects that are a result of systemic muscarinic receptor blockade. Medications are successful for many patients but compliance is poor and many patients discontinue the medications as a result of side effects, cost, and insufficient symptom improvement.

Percutaneous tibial nerve stimulation (PTNS) is a newer treatment modality that provides neuromodulation to the pelvic floor by stimulating the posterior tibial nerve. This nerve is accessed with a fine needle electrode that is inserted in the medial portion of the ankle. This area has long been recognized as having nerve projections to the sacral nerve plexus and can modulate bladder activity. Several studies have clearly demonstrated the effectiveness of neuromodulation to treat urge incontinence.

There have been studies comparing the efficacy of pharmacotherapy versus PTNS. In one study, 49% of subjects taking fesoterodine fumarate for urge incontinence reported an improvement in symptoms of overactive bladder. In other studies, 79.5% of patients undergoing PTNS reported improvement or cure. Although studies report similar improvement or cure between the two treatment modalities, there is no evidence of the efficacy of using both PTNS and pharmacotherapy concurrently. This study is aimed at proving synergy between the two treatment modalities when used together in an effort to administer smaller doses of anticholinergic agents, while obtaining comparable or improved urge incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Female ages > 18 and < 100 years old without childbearing potential
* History of overactive bladder

  * with or without urge incontinence)
  * with or without a history of previous anticholinergic use
* At least 8 voids per 24 hours documented by history and physical and voiding diary

Exclusion Criteria:

* Has had PTNS modulation in the past
* Has a primary complaint of stress urinary incontinence
* History of an allergy or sensitivity to tolterodine tartrate tablets or its ingredients
* History of an allergy or sensitivity to fesoterodine tartrate tablets or its ingredients
* Has a recent positive urinalysis for infection
* Has taken anticholinergic medication in the last 4 weeks for overactive bladder
* Has any of the following:

  * pacemakers or implantable defibrillators
  * excessive bleeding
  * urinary or gastric retention
  * nerve damage and/or neuropathy
  * myasthenia gravis, uncontrolled narrow angle glaucoma
  * liver disease or kidney disease
  * QT prolongation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Cornella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona (MCSB and MCH), Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo: Participants were to be given PTNS + 4mg of fesoterodine fumarate (12 weeks), Washout (4 weeks), PTNS + placebo (12 weeks)
- PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate: Participants were to be given PTNS + placebo (12 weeks), washout (4 weeks), PTNS + 4mg of fesoterodine fumarate (12 weeks)
Period: First Intervention
Arm/Group | PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo | PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Washout Period of 4 Weeks
Arm/Group | PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo | PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Study Terminated | 2 | 1
Period: Second Intervention
Arm/Group | PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo | PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo | PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Urinary Voids Per 24 Hours After 12 Weeks of Therapy
Time Frame: From baseline to 12 weeks post treatment
Population: The study was terminated due to a low recruitment rate prior to subjects completing treatment.
Groups:
- PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo: Participants were to be given PTNS + 4mg of fesoterodine fumarate first for 12 weeks, and followed by 4 weeks of washout followed by 12 weeks of PTNS + placebo
- PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate: Participants were to be given PTNS + placebo for 12 weeks followed by 4 weeks of washout followed by 12 weeks of PTNS + 4mg of fesoterodine fumarate
Arm/Group | PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo | PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mean Change in Urinary Urge Incontinence Episodes in 24 Hours
Time Frame: Baseline, 12 weeks post treatment
Population: The study was terminated due to a low recruitment rate prior to subjects completing treatment.
Arm/Group | PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo | PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Voids Causing Waking
Time Frame: From baseline to 12 weeks post treatment
Population: The study was terminated due to a low recruitment rate prior to subjects completing treatment.
Arm/Group | PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo | PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Volume Voided Per Day
Time Frame: From baseline to 12 weeks post treatment
Population: The study was terminated due to a low recruitment rate prior to subjects completing treatment.
Arm/Group | PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo | PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Urgency Episodes Scored by the Indevus Urgency Severity Scale (IUSS)
Description: The IUSS has 4 levels: none, mild, moderate, and severe. An episode characterized as severe according to this scale would qualify as an urgency episode.
Time Frame: baseline, 12 weeks post treatment
Population: The study was terminated due to a low recruitment rate prior to subjects completing treatment.
Arm/Group | PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo | PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Score on Overactive Bladder Questionnaire (QAB-q)
Description: The QAB-q is a self-administered, 33-item questionnaire containing a symptom bother and health related quality of life scale. Each item has a choice of 6 responses, ranging from "not at all" to "a very great deal." Therefore, the total score could range from 33 (no discomfort) to 198 (great discomfort).
Time Frame: Baseline, 12 weeks post treatment
Population: The study was terminated due to a low recruitment rate prior to subjects completing treatment.
Arm/Group | PTNS + Fesoterodine Fumarate First, Then PTNS + Placebo | PTNS + Placebo First, Then PTNS + Fesoterodine Fumarate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- While on PTNS + Fesoterodine Fumarate First: Participants were given PTNS + 4mg of fesoterodine fumarate (12 weeks)
- While on PTNS + Placebo First: Participants were given PTNS + placebo (12 weeks)
- While on PTNS + Placebo Second: Participants were to be given PTNS + placebo (12 weeks)
- While on PTNS + Fesoterodine Fumarate Second: Participants were to be given PTNS + 4mg of fesoterodine fumarate (12 weeks)
Arm/Group | While on PTNS + Fesoterodine Fumarate First | While on PTNS + Placebo First | While on PTNS + Placebo Second | While on PTNS + Fesoterodine Fumarate Second
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | While on PTNS + Fesoterodine Fumarate First (N=2) | While on PTNS + Placebo First (N=2) | While on PTNS + Placebo Second (N=0) | While on PTNS + Fesoterodine Fumarate Second (N=0)
Irregular heartbeat/palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Subject was having irregular heartbeat/palpitations and this is a potential side effect of Toviaz (study drug). However, after the blind was broken, it was determined that she was taking the placebo, so palpitations were not due to the Toviaz.

LIMITATIONS AND CAVEATS:
The study was terminated due to a low recruitment rate prior to subjects completing treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No